CLINICAL TRIAL: NCT00269529
Title: Postoperative Analgesia After Total Knee Arthroplasty. A Comparison of Continuous Femoral Block and Extensive Intraoperative Infiltration With Local Anesthetic Supplemented With Intraarticular Bolus the Following Day.
Brief Title: Intraarticular Analgesia After Total Knee Arthroplasty, a Randomised Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other); Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050003
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: postoperative pain; knee arthroplasty; analgesia; infiltration; femoral nerve block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

INTERVENTIONS:
Procedure: femoral nerve block
Procedure: knee infiltration and injection via catheter

SUMMARY:
The study aims to compare two different kinds of pain treatment after total knee replacement (operation with artificial knee joint): 1) a large local injection in and around the knee, supplemented with injection the day after, or 2) the department's conventional pain treatment consisting of continuous nerve block in the groin.

DETAILED DESCRIPTION:
Postoperative pain after total knee arthroplasty is moderate to severe and can be difficult to treat. The current use of femoral nerve block by ropivacain pump for 48 hours provides considerable analgesia, but patients often experience slight motor block, inhibiting rehabilitation, and pain in the posterior part of the knee, innervated by the sciatic nerve. This study compares femoral nerve block to a new technique, where ropivacaine, ketorolac and adrenalin is used to infiltrate the tissue in and around the knee joint during surgery, and is injected by an intraarticular catheter at 10 pm on the day of surgery and again at 10 am the day after. Data of pain scores, analgesia consumption, adverse effects and mobilisation is collected for the first four postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for primary total knee arthroplasty due to primary arthrosis

Exclusion Criteria:

* Patients unable to provide informed consent
* patients with contraindications for spinal anesthesia
* patients with known hypersensitivity towards the used drugs
* patients with severe chronic neurogenic pain or sensitivity disorders in the leg to be operated
* patients who have undergone major bone surgery in the knee to be operated

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2005-02; Study Completion 2006-03

PRIMARY OUTCOMES:
pain, by numeric rating scale
pain, by consumption of analgesics
side effects
return of function

CONTACTS AND LOCATIONS:
Overall Officials: Else Tønnesen, Professor, Principal Investigator — Department of Anesthesiology, Aarhus University Hospital, Aarhus, Denmark; Kjeld Søballe, Professor, Principal Investigator — Orthopedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Aarhus Hospital, Tage Hansens Gade, Aarhus, Denmark